CLINICAL TRIAL: NCT00788827
Title: A Phase I Safety and Tolerability Study Following the Infusion of Autologous Expanded Progeny of an Adult CD34+ Stem Cell Subset (InsulinCytes) to Patients With Type I Diabetes Mellitus and a Successful Renal Transplant
Brief Title: Autologous Adult Stem Cells to Patients With Type 1 Diabetes and a Successful Renal Transplant
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HHSC 005; CRO0472 (Other: Imperial College London)
Record Dates: First submitted 2008-11-10; First posted 2008-11-11 (Estimated); Results first posted 2019-11-18 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-10

CONDITIONS: Type 1 Diabetes; Type 2 Diabetes
Keywords: diabetes type I; diabetes type 2; renal transplant; stem cells; successful renal transplant
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Autologous stem cells
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Autologous CD34+ stem cells (Experimental): Up to 5 x 10 log 8 of autologous stem cells on a single occasion
  Interventions: Biological: Autologous CD34+ stem cells

INTERVENTIONS:
Biological: Autologous CD34+ stem cells — Up to 5 x 10 log 8 of autologous stem cells on a single occasion

SUMMARY:
This is a phase I study to assess the safety and tolerability of infusing expanded stem cells into the pancreas of patients with type I diabetes and a successful renal transplant. The stem cells used in this study occur naturally in the body and are collected from each recipient by a procedure called leukapheresis. The cells are then expanded and differentiated into insulin-like cells in a sterile suite before being injected into the body or tail of the pancreas of the recipient.

DETAILED DESCRIPTION:
Islet transplantation as a potential treatment for diabetes has been investigated extensively over the past 10 years. Such an approach, however, will always be limited mainly because it is difficult to obtain sufficiently large numbers of purified islets from cadaveric donors. One alternative to organ or tissue transplantation is to use a renewable source of cells. Adult stem cells are clonogenic cells capable of both self-renewal and multilineage differentiation. These cells have the potential to proliferate and differentiate into any type of cell and to be genetically modified in vitro, thus providing cells, which can be isolated and used for transplantation.

Recent studies have given well-defined differentiation protocols, which can be used to guide stem cells into specific cell lineages as neurons, cardiomyocytes and insulin-secreting cells. Moreover, these derived cells have been useful in different animal models. In this regard, insulin-secreting cells derived from R1 mouse embryonic stem cells restore blood glucose concentrations to normal when they are transplanted into streptozotocin-induced diabetic animals. Our group has isolated stem cells (Cluster Designated (CD) 34 positive subset of stem cells) that are capable of differentiating into multiple tissue types ex vivo. In defined conditions, in culture, about 40 percent of the cells produce insulin and reduce blood sugar levels in streptozotocin-induced mice.

Clinically, we have performed a phase I trial of stem cell administration to patients with liver insufficiency. The procedure was well tolerated with no specific side effects and with sustained signs of clinical benefit. These results support this protocol for the application of adult stem cell therapy in the treatment of diabetes.

In order to evaluate potential clinical applications for these recent advances we have designed a prospective Phase I clinical study of the expanded progeny of an adult CD34 positive subset (InsulinCytes) injected directly into the body and tail of the pancreas of the participants via selective catheterisation of the splenic artery. The study group consists of patients with complicated diabetes mellitus type I plus kidney transplantation with the aim of ascertaining whether this confers clinical benefit as a treatment model for diabetes.

Granulocyte colony-stimulating factor (G-CSF) will be administered to suitable patients to mobilise their haematopoietic stem cells (HSCs) from the bone marrow into the peripheral circulation. These blood cells will be collected from each patient by leukapheresis. CD34 positive stem cells will then be isolated by immunoselection and introduced into a Nunc cell factory where the subset of CD34 positive stem cells will be allowed to attach to the plastic trays within the cell factory for 2 hours at 37 degrees C in 5 percent carbon dioxide. After this period the non-attached CD34 positive cells will be washed from the system and the progeny of the attached cells secreted into the supernatant media expanded in the presence of growth medium supplemented with growth factors. At the end of 6 days expansion, the stem cells will be differentiated into insulin and c-peptide protein excreting cells over the next 14 days by the addition of specified reagents/growth factors and continued incubation at 37 degrees C in 5 percent carbon dioxide in accordance with the principles of Good Manufacturing Practice (GMP). As an optional step the cells can be labelled with iron oxide to allow tracking of the cells by Magnetic Resonance Imaging (MRI) scan, before being infused into the patient.

An ongoing institute experience with liver failure patients who have been infused with undifferentiated stem cells has shown that an administered dose of up to 2 x 10 log 9 cells was well tolerated. The proposed study group will consist of 10 Type I or Type 2 diabetic patients who have had a successful previous kidney transplant.

The primary purpose of the study is to assess the safety and tolerance of stem cell infusion into the pancreas and then to assess the impact of this new modality in the treatment of diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged from 16 to 65 years of age
* Patient with Type I or Type 2 diabetes mellitus plus:
* Successful previous kidney transplant.
* Good kidney allograft function /no episodes of rejection for at least one year post-transplant
* Not taking steroids as part of standard immuno-suppression
* Has a WHO performance score of less than 2
* Has a life expectancy of at least 3 months
* Ability to give written consent
* Women of childbearing potential may be included, but must use a reliable and appropriate contraceptive method

Exclusion Criteria:

* Patients below the age of 16 or above the age of 65 years
* Patients with chronic pancreatitis and poor exocrine pancreatic function
* Pregnant or lactating women
* Patients with recent recurrent GI bleeding or spontaneous bacterial peritonitis
* Patients with evidence of HIV or other life threatening infection
* Patients unable to give written consent
* Patients with a history of hypersensitivity to G-CSF
* Patients who have been included in any other clinical trial within the previous month

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2008-11 (Actual); Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Pusey, MD, Principal Investigator — Imperial College London
Locations (1):
- Imperial College NHS Healthcare Trust, Hammersmith Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Autologous CD34+ Stem Cells
Started | 7
Completed | 5
Not Completed | 2
Not completed — Lack of Efficacy | 2

BASELINE CHARACTERISTICS:
Groups:
- Single Arm: Autologous CD34+ Stem Cells
Arm/Group | Single Arm
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.6 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Adverse Events
Description: Safety will be evaluated in terms of adverse events graded according to CTCTAE toxicity criteria and laboratory test results. All adverse events will also be graded for relationship to treatment and as expected and unexpected.
Time Frame: 14 days
Measure: Number; unit: participants
Groups:
- Autologous Stem Cells: Up to 5 x 10 log 8 of autologous stem cells on a single occasion
  Autologous CD34+ stem cells: Up to 5 x 10 log 8 of autologous stem cells on a single occasion
Arm/Group | Autologous Stem Cells
Number analyzed (Participants) | 7
participants
  Haematoma at femoral catheter insertion | 1
  Fatigue | 7

2. Secondary Outcome: Hba1C Data of Pre and Post Stem Cell Infusion
Description: Mean HbA1c laboratory measurements pre and post stem cell infusion
Time Frame: 12 weeks
Population: Patients who were infused with stem cells
Measure: Mean (Standard Deviation); unit: percentage
Groups:
- Pre Infusion of Stem Cells: Before the infusion of stem cells
- Post Infusion of Stem Cells: After the infusion of stem cells
Arm/Group | Pre Infusion of Stem Cells | Post Infusion of Stem Cells
Number analyzed (Participants) | 5 | 5
percentage | 7.2 (1.3) | 7.24 (1.2)
Statistical Analysis 1: Comparison: Pre Infusion of Stem Cells vs Post Infusion of Stem Cells; Each participants Hba1c (%) lab result was analysed pre and post stem cell infusion to achieve 2 mean readings per participant; Test type: Other; p < 0.05, Mixed Models Analysis

3. Secondary Outcome: Insulin Level
Description: Mean insulin requirement was calculated for each participant pre and post stem cell infusion
Time Frame: 12 weeks
Population: Participants who received a stem cell infusion
Measure: Mean (Standard Deviation); unit: iu/day
Arm/Group | Pre Infusion of Stem Cells | Post Infusion of Stem Cells
Number analyzed (Participants) | 5 | 5
iu/day | 59.4 (25.7) | 54.06 (18.2)

4. Secondary Outcome: Amylase Level
Description: Each participant had mean amylase data analysed to give a pre and post mean result
Time Frame: 12 weeks
Population: Participants who received a stem cell infusion
Measure: Mean (Standard Deviation); unit: units/L
Arm/Group | Pre Infusion of Stem Cells | Post Infusion of Stem Cells
Number analyzed (Participants) | 5 | 5
units/L | 48.49 (25.2) | 75.52 (34.2)

5. Secondary Outcome: Serum Creatinine
Description: Each participant had serum creatinine analysis pre and post stem cell infusion to give mean result
Time Frame: 12 weeks
Population: Participants who received stem cell infusion
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Pre Infusion of Stem Cells | Post Infusion of Stem Cells
Number analyzed (Participants) | 5 | 5
umol/L | 128.22 (11.9) | 118.64 (15.5)

ADVERSE EVENTS:
Time Frame: 12 weeks
Groups:
- Single Arm: Autologous stem cells
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 7/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=7)
Fatigue (Nervous system disorders) | 7 (7)
Haemotoma (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes